CLINICAL TRIAL: NCT05179967
Title: Guo's visceRal artEries Reconstruction :The Prospective, Multiple Center, Objective Performance Criteria Clinical Trial About the sAfTy and Efficacy of WeFlow-JAAATM Stent Graft System.(GREAT Study)
Brief Title: Safety and Efficacy Study of WeFlow-JAAA Stent Graft System for Complex Abdominal Aortic Aneurysm(GREAT Study)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hangzhou Endonom Medtech Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: WEIQIANG202101
Record Dates: First submitted 2021-12-17; First posted 2022-01-06 (Actual); Last update posted 2022-03-16 (Actual); Status verified 2022-03

CONDITIONS: Juxtarenal Abdominal Aortic Aneurysm

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- WeFlow-JAAA Stent Graft System (Experimental)
  Interventions: Device: WeFlow-JAAA Stent Graft System

INTERVENTIONS:
Device: WeFlow-JAAA Stent Graft System — WeFlow-JAAA Stent Graft System consists of abdominal main body of inner embedded stent graft , abdominal main bifurcation stent graft, extension stent graft and branch stent graft. The abdominal main body of inner embedded stent graft is composed of abdominal main embedded covered stent and conveyor, the abdominal main bifurcated stent graft is composed of abdominal main bifurcated stent and conveyor, the extended stent is composed of extended stent graft and conveyor, and the branch vascular stent graft is composed of branch vascular stent and conveyor. The abdominal main body of inner embedded stent graft, abdominal main bifurcation stent graft, extension stent graft and branch vascular stent graft are pre-installed in the corresponding conveyor respectively.

SUMMARY:
A prospective, multi-center, objective performance criteria clinical trial to evaluate the safety and efficacy of WeFlow-JAAA stent graft system manufactured by Hangzhou Endonom Medtech Co., Ltd. for the complex abdominal aortic aneurysm.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-80 years old, regardless of gender;
2. Subjects who were diagnosed with Juxtarenal and Pararenal abdominal aortic aneurysms and needed to reconstruct the blood supply of superior mesenteric artery and bilateral renal arteries;
3. Have appropriate vascular conditions, mainly including:

   * The distance between the upper edge of the aneurysm and the lower edge of the opening of superior mesenteric artery ≥ 4mm;
   * The angle between the proximal aneurysm neck and the aortic long axis near the opening of superior mesenteric artery ≤ 60 ° ;
   * The aortic diameter at the opening of superior mesenteric artery ranges from 18 to 34 mm ；
   * The diameter range of the starting part of superior mesenteric artery is 5-12mm；
   * The diameter range of the initial part of bilateral renal arteries is 4.5-10mm;
   * Length of non bifurcated segment of superior mesenteric artery and renal artery ≥ 10mm;
   * Blood vessel diameter at the bifurcation of abdominal aorta ≥ 16mm；
   * The length of distal anchoring area of iliac artery ≥ 15mm;
   * The diameter range of distal anchoring area of iliac artery is 8-24mm;
   * With appropriate femoral artery、iliac artery and upper limb artery approaches, endovascular treatment can be performed.
4. Those who can understand the purpose of the trial, voluntarily participate in the study, sign the informed consent form by themselves or their legal representative, and are willing to complete the follow-up according to the protocol requirements.

Exclusion Criteria:

1. Patients with ruptured abdominal aortic aneurysm, pseudoaortic aneurysm and dissecting aortic aneurysm with hemodynamic instability;
2. Infectious aortic disease, Takayasu arteritis, Marfan syndrome (or other connective tissue diseases);
3. Severe stenosis, calcification and mural thrombosis in the proximal anchoring area of the stent;
4. Other vascular diseases need to be intervened in the same operation (such as coronary artery and carotid artery) and the postoperative drug treatment scheme is affected;
5. There is a history of myocardial infarction, TIA or cerebral infarction in recent 3 months;
6. The subject has a history of abdominal aortic surgery or endovascular repair;
7. Patients with severe liver, kidney, lung and cardiac dysfunction before operation [subjects with serum creatinine level > 150umol / L; alanine aminotransferase (ALT) or aspartate aminotransferase (AST) exceeds 5 times the upper normal limit; total serum bilirubin (STB) subjects who exceed 2 times the upper limit of normal; subjects whose left ventricular ejection fraction is less than 50% by color Doppler echocardiography.];
8. Patients with acute systemic infection;
9. Patients with contraindications to antiplatelet agents and anticoagulants;
10. Subjects are allergic to contrast agents, anesthetics, stents and conveyor materials;
11. Subjects cannot tolerate anesthesia;
12. Subjects Women who are pregnant or lactating or who cannot use contraception during the trial;
13. Subjects whose life expectancy is less than 12 months (such as advanced malignant tumor);
14. Subjects have participated in clinical trials of other drugs or devices in the same period;
15. The researchers determine that the subjects' vascular conditions affect the revascularization of branch arteries or are combined with other diseases and are not suitable to participate in this study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Estimated)
Dates: Start 2022-02-23 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Rate of no major adverse events occurred within 30 days after operation | Within 30th day after operation
  The main adverse events within 30 days after operation refer to all-cause death, myocardial infarction, renal failure, respiratory failure, ischemic stroke, intestinal necrosis, severe ischemia or necrosis of lower limbs and paraplegia within 30 days after operation. Among them, renal failure leads to lasting dialysis, renal transplantation or other fatal results. Respiratory failure leads to significantly prolonged intubation time, tracheotomy, deterioration of pulmonary function or other fatal results. Intestinal necrosis refers to intestinal ischemia that requires intestinal resection or leads to other fatal results. Severe ischemia of lower limbs refers to new severe claudication or resting pain after operation.
The success rate of treatment of abdominal aortic aneurysm 12 months after operation | 12 months after operation
  Immediate postoperative technical success refers to the successful delivery of the conveyor of aortic and branch covered stents to the predetermined position, the accurate positioning and successful deployment of the stent, and the conveyor can be safely withdrawn from the body. At the end of the operation, there is no type I and III internal leakage and the branch stent is unobstructed.

SECONDARY OUTCOMES:
Rate of all cause mortality | Before discharge, 30 days, 6 months, 12 months and 2-5 years after operation
  All cause death refers to death from any cause during the follow-up period
Rate of abdominal aortic aneurysm related mortality | Before discharge, 30 days, 6 months, 12 months and 2-5 years after operation
  Rate of abdominal aortic aneurysm related death refers to death caused by aneurysm rupture or surgery for aortic aneurysm
Incidence of serious adverse events | Before discharge, 30 days, 6 months, 12 months and 2-5 years after operation
  Serious adverse events refer to events that lead to death or serious deterioration of health status during clinical trials, including fatal diseases or injuries, permanent defects in body structure or function, and the need for medical or surgical intervention to avoid permanent defects in body structure or function.
Incidence of device related adverse events | Before discharge, 30 days, 6 months, 12 months and 2-5 years after operation
  Device related adverse events refer to adverse medical events related to the use of devices during clinical trials. However, normal postoperative stress reactions, such as fever and chest and back discomfort, should be distinguished. If they are judged as normal postoperative stress reactions by the researchers, they need not be recorded in adverse events. Recording device related adverse events refers to the situation that the investigator determines to be definitely related, possibly related or unable to determine with the test device.
Incidence of type I or type III internal leakage | Intraoperative, before discharge, 6 months, 12 months
  The internal leakage shown by DSA or CTA was recorded. The internal leakage occurred during the operation and the adjuvant treatment is not recorded. Internal leakage after operation and untreated internal leakage in the same subject at different follow-up stages shall be calculated once.
Incidence of aortic covered stent displacement | 6 and 12 months after operation
  CTA was observed and recorded 6 months and 12 months after operation to check whether the stent was displaced. The main stent and branch stent were recorded and evaluated. Displacement was defined as the displacement of aortic and branch covered stents at the postoperative follow-up node more than 10mm compared with that before discharge.
Patency rate of postoperative branches | Before discharge, 6 months, 12 months
  CTA was observed and recorded before discharge, 6 months and 12 months to evaluate the revascularization of branches of renal artery and superior mesenteric artery, and whether there was occlusion, stenosis or stent thrombosis. Postoperative branch vessel stenosis ≤ 50% is regarded as unobstructed.
Incidence of conversion to open surgery or secondary interventional surgery for abdominal aortic aneurysm | Before discharge, 6 months, 12 months, 2 ~ 5 years
  To evaluate whether the subjects were converted to open surgery or secondary interventional surgery due to abdominal aortic aneurysm.

CONTACTS AND LOCATIONS:
Locations (1):
- The General Hospital of the People's Liberation Army, Beijing, China